CLINICAL TRIAL: NCT02106013
Title: Association Between HDL Functions and Atherosclerotic Burden in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Professor of Cardiology, University of Campinas, Brazil
Other Study IDs: BHS2
Record Dates: First submitted 2014-03-30; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Low HDL Cholesterol
Keywords: HDL; Carotid artery intima-media thickness; Cholesterol efflux capacity; Antioxidant effect of HDL; Susceptibility to oxidation of HDL; Anti-inflammatory effect of HDL; Platelet aggregation inhibition by HDL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low HDL-C: Study participants with HDL-C levels below the 10th percentile (HDL-C ≤32 mg/dL)
- Intermediate HDL-C: Study participants with HDL-C levels between 40th and 60th percentiles (40≤HDL-C≤67 mg/dL)
- High HDL-C: Study participants with HDL-C levels above the 90th percentile (HDL-C ≥78mg/dL)

SUMMARY:
This is a study of HDL function in healthy individuals classified in three groups according to their HDL-cholesterol levels (Low HDL-C, Intermediate HDl-C and High HDL-C), with the purpose of investigating which characteristics of the HDL particle might be associated to atherosclerotic burden, characterized by carotid intima-media thickness above 1mm.

DETAILED DESCRIPTION:
Selection: Study participants are initially selected trough the evaluation of consecutive lipid profiles from individuals who spontaneously seek governmental primary care centers of the city of Campinas, Sao Paulo, Brazil. Telephone-based screening interviews are performed, followed by in-person clinical evaluation and blood exams.

Biochemical analyses: Glucose, triglycerides, HDL-C and c-reactive protein (CRP) are measured in an automated Modular® Analytics Evo (Roche Diagnostics, Burgess Hill, West Sussex, UK), using Roche Diagnostics® reagents (Mannheim, Germany). LDL-cholesterol is calculated by the Friedewald formula. Serum insulin levels are measured using ELISA (Millipore, Massachusetts, USA). The Homeostasis Model Assessment (HOMA) Calculator version 2.2 (University of Oxford, UK) is used to estimate insulin sensitivity. Apolipoproteins A-I and B-100 and lipoprotein (a) are determined by nephelometry in an automated system and reagents from Dade-Behring® (Marburg, Germany).

Carotid artery ultrasound: Carotid artery atherosclerosis is estimated by using high-resolution B-mode ultrasound, at the posterior wall of the common carotid artery.

Lipoprotein isolation: HDL from each study participant is isolated from plasma, through ultracentrifugation (Beckman Coulter Inc., Palo Alto, USA).

HDL chemical composition: Using commercially available enzymatic kits, HDL content of total proteins, total cholesterol, free cholesterol, phospholipids, triglycerides and apolipoprotein A-I are measured. Cholesteryl ester (CE) is calculated as the difference between total cholesterol and free cholesterol times 1.67. HDL molar concentration is estimated based on particle total mass and molecular weight.

HDL physical-chemical characterization: HDL particle size is determined using dynamic light scattering, and zeta potential using laser Doppler micro-electrophoresis.

Determination of proteins involved in HDL metabolism: Cholesteryl ester transfer protein, phospholipids transfer protein, lipoprotein lipase, hepatic lipase and lecithin:cholesterol acyl transferase activities are determined trough radiometric exogenous assays.

HDL functions: Cholesterol efflux capacity, antioxidant activity, susceptibility to oxidation, anti-inflammatory activity and platelet aggregation inhibition are measured using straightforward and consolidated methodologies.

Statistical Analyses: Differences between groups are evaluated using ANOVA or Kruskal-Wallis, with Bonferroni's post-hoc multiple comparison analysis, according to variable distribution. Chi-Square is used to compare categorical data. Analysis of covariance (ANCOVA) adjusted for confounding variables is also used, after checking variables with histograms, normality plots, and residual scatter plots that tested for linearity, normality, and variance. Pearson's correlation test is used to assess the relationships between variables. A two-sided p-value of 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* glucose <100 mg/dL
* Urea <71 mg/dL
* Creatinine < 1.20 mg/dL
* Uric acid <7.0 mg/dL
* Alanine aminotransferase <50 U/L
* Aspartate aminotransferase < 33 U/L
* Gamma-glutamyl transferase <71 U/L
* Alkaline phosphatase <129 U/L
* Thyroid stimulating hormone between 0.41 and 4.50 μUI/mL
* Free thyroxin between 0.9 and 1.8 ng/dL

Exclusion Criteria:

* Symptomatic cardiovascular disease
* LDL-cholesterol ≥130 mg/dL
* Triglycerides ≥150 mg/dL
* Metabolic syndrome
* BMI ≥ 30 kg/m2
* Smoking habit
* Daily intake of alcohol >14g
* Regular use of medical treatments

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who sought governmental primary care centers of the city of Campinas, SP, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-04; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cholesterol efflux capacity of HDL | The analysis will be performed using plasma obtained at admission into the study
  This is a cross-sectional study and as such the cholesterol efflux capacity will be measured using the plasma sample collected at admission into the study

SECONDARY OUTCOMES:
Antioxidant activity of HDL | The analysis will be performed using plasma obtained at admission into the study
  This is a cross-sectional study and as such the cholesterol efflux capacity will be measured using the plasma sample collected at admission into the study
Susceptibility to oxidation of HDL | The analysis will be performed using plasma obtained at admission into the study
  This is a cross-sectional study and as such the cholesterol efflux capacity will be measured using the plasma sample collected at admission into the study
Anti-inflammatory activity of HDL | The analysis will be performed using plasma obtained at admission into the study
  This is a cross-sectional study and as such the cholesterol efflux capacity will be measured using the plasma sample collected at admission into the study
Platelet aggregation inhibition by HDL | The analysis will be performed using plasma obtained at admission into the study
  This is a cross-sectional study and as such the cholesterol efflux capacity will be measured using the plasma sample collected at admission into the study

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, PhD MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil